CLINICAL TRIAL: NCT06228196
Title: Cohort Study of Clinical and Neuroimaging Characteristics for BPPV Patients in China
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-566
Record Dates: First submitted 2024-01-08; First posted 2024-01-29 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: BPPV; Vertigo; Vertigo, Peripheral
Keywords: BPPV; residual dizziness; Vertigo; Neuroimaging; Epidemic
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPPV patients: Confirmed diagnosis of BPPV
  Interventions: Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum
- Healthy controls: Healthy subjects who have not had BPPV
  Interventions: Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum

INTERVENTIONS:
Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum — Simultaneous cortico-spinal magnetic resonance imaging data were collected in a strong magnetic field and collected the serum of participants.

SUMMARY:
The main objective is to analyze the abnormality of physical condition, mental health and blood examination of the patients with benign paroxysmal positional vertigo (BPPV). Besides, the investigators aim to establish a database of BPPV based on multimodal magnetic resonance imaging data in the brain to identify high-risk patients with residual dizziness (RD) and systematically establish the comprehensive assessment system for the precise diagnosis, treatment and recovery of RD, optimize the tactics of BPPV management in China.

DETAILED DESCRIPTION:
This is an observational, longitudinal, and single-center study. Confirmed BPPV cases will complete the following programs before and after 1 and 6 months of treatment for exploring biological mechanism and predictive biomarkers of BPPV: 1) fill in the behavioral psychological scales, 2) submit blood samples at a local laboratory, 3) receive 3 times brain MRI scan. The healthy controls will complete the same programs as BPPV-group mentioned above only at the time of inclusion. The investigators will establish the brain MRI database containing neuropsychological scales and blood parameters of BPPV in China.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of BPPV/Healthy subjects who have not had BPPV

Exclusion Criteria:

* History of organic diseases in central nervous system and mental disorder, such as tumors, infections, depressive disorder, schizophrenia, etc. Claustrophobic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be carried out in the First Affiliated Hospital Xi'an Jiaotong University for patients who had diagnosis of BPPV by the Dix-Hallpike maneuver or Supine Roll test.
  The healthy control population will be searched in the primary care services, media and social networks.
  All participants will sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences between patients with BPPV and control group in brain structure | baseline and 1 and 6 months
  The changes of brain volume (mm3) are evaluated by structural MRI
Differences between two groups in brain function | baseline and 1 and 6 months
  The changes of brain functional connectivity intensity are evaluated by functional MRI
Changes on vertigo symptoms | baseline and 1 and 6 months
  Vertigo is assessed with the Dizziness Handicap Inventory (DHI Scale)
Changes on vertigo symptoms | baseline and 1 and 6 months
  Vertigo is also assessed with the Activities-specific Balance Confidence Scale (ABC Scale)
Changes on vertigo symptoms | baseline and 1 and 6 months
  Vertigo is also assessed with the Visual Vertigo Analogue Scale (VVAS)
Difference in blood markers between the two groups | baseline and 1 and 6 months
  All subjects underwent fasting vein blood collection of about 5 ml at about 8 a.m. Blood indices related to BPPV and related clinical symptoms were screened, the inflammatory index is interleukin-6（IL-6）
Difference in blood markers between the two groups | baseline and 1 and 6 months
  Immunology-related index in the blood sample is superoxide dismutase (SOD)
Difference in blood markers between the two groups | baseline and 1 and 6 months
  Inflammatory index in the blood sample is neutrophils/lymphocytes

SECONDARY OUTCOMES:
Differences in Fatigue between the two groups | baseline and 1 and 6 months
  Fatigue is assessed with the Multidimensional Fatigue Inventory (MFI). A higher score represents a worse outcome. The MFI is a 20-item self-report instrument covering four dimensions (general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity) designed to measure fatigue.
Differences in Sleep between the two groups | baseline and 1 and 6 months
  Sleep quality is assessed with Pittsburgh Sleep Quality Index (PSQI). A higher score corresponding to a worse sleep quality.
Differences in cognition between the two groups | baseline and 1 and 6 months
  The cognition is assessed with Montreal Cognitive Assessment (MoCA). Higher scores (0-30) are related to a better performance.
Differences in executive function between the two groups | baseline and 1 and 6 months
  The executive function is assessed with Trail Making Test A and B. Participants are asked to connect sequential numbers (TMT-A) and interconnect sequential numbers and letters (TMT-B).
Difference in anxiety between the two groups | baseline and 1 and 6 months
  Anxiety is assessed with Beck Anxiety Inventory (BAI). A higher score corresponding to more severe anxiety symptoms.
Difference in depression between the two groups | baseline and 1 and 6 months
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9). A higher score corresponding to more severe depression symptoms.
Differences in verbal memory and working memory between the two groups | baseline and 1 and 6 months
  Verbal memory is assessed with the Auditory Verbal Learning Test (AVLT). A 12-word list are read by examiner three times and participants are asked to recall them followed by each presentation, which was called "immediate recall". The "short delayed recall" and "long delayed recall" ask the participants to recall the above 12-word list 5 minutes and 20 minutes later, the correctly recalled number of words are recorded. Finally, the subjects are instructed to recognize the learned words from a 24-words list which consisted of above learned 12-words list and a new unlearned 12-words list. Working memory is assessed with the Digit Span Backward. Participants are asked to repeat the numbers in the reverse order the examiner read them aloud and a higher score corresponding to a better outcome.
Differences in auditory attention between the two groups | baseline and 1 and 6 months
  Auditory attention is assessed with the Digit Span Forward. Participants are asked to repeat the numbers in the order the examiner read them aloud and a higher score corresponding to a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wang, M.D., Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China